CLINICAL TRIAL: NCT01322594
Title: A Phase 1, Single Ascending Dose Study to Evaluate the Safety of MEDI2338 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Safety of MEDI2338 in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CD-RI-MEDI2338-1033; 2010-022879-54 (EudraCT Number)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- MEDI2338 10 MG (Experimental): MEDI2338 (10 mg) administered as a single, fixed intravenous (IV) dose over a minimum of 60 minutes using an infusion pump
  Interventions: Biological: MEDI2338
- MEDI2338 30 MG (Experimental): MEDI2338 (30 mg) administered as a single, fixed IV dose over a minimum of 60 minutes using an infusion pump
  Interventions: Biological: MEDI2338
- MEDI2338 100 MG (Experimental): MEDI2338 (100 mg) administered as a single, fixed IV dose over a minimum of 60 minutes using an infusion pump
  Interventions: Biological: MEDI2338
- MEDI2338 300 MG (Experimental): MEDI2338 (300 mg) administered as a single, fixed IV dose over a minimum of 60 minutes using an infusion pump
  Interventions: Biological: MEDI2338
- MEDI2338 1000 MG (Experimental): MEDI2338 (1000 mg) administered as a single, fixed IV dose over a minimum of 60 minutes using an infusion pump
  Interventions: Biological: MEDI2338
- Placebo (Placebo Comparator): Placebo administered as a single, fixed IV dose over a minimum of 60 minutes using an infusion pump
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI2338 — MEDI2338 single intravenous (IV) dose (lowest dose)
  Arms: MEDI2338 10 MG
Biological: MEDI2338 — MEDI2338 single IV dose (next highest dose)
  Arms: MEDI2338 30 MG
Biological: MEDI2338 — MEDI2338 single IV dose (next highest dose)
  Arms: MEDI2338 100 MG
Biological: MEDI2338 — MEDI2338 single IV dose (next highest dose)
  Arms: MEDI2338 300 MG
Biological: MEDI2338 — MEDI2338 single IV dose (highest dose)
  Arms: MEDI2338 1000 MG
Other: Placebo — Placebo single IV dose
  Arms: Placebo

SUMMARY:
Phase I study to evaluate the safety and tolerability of single ascending intravenous doses of MEDI2338 in subjects with stable, mild to moderate chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 40 years at time of screening.
* Females of non-childbearing potential defined as surgically sterile or at least 2 years postmenopausal.
* Males, unless surgically sterile, must use 2 highly effective methods of birth control from screening through end of trial.
* A diagnosis of mild to moderate COPD.
* Cigarette smoking history of ≥10 pack years.
* Ability to understand and comply with protocol requirements, instructions and restrictions.
* COPD symptoms adequately controlled on a therapeutic regimen that has not changed in the 4 weeks prior to screening.

Exclusion Criteria:

* Current diagnosis of any respiratory condition other than COPD.
* Active or history of any disease or condition that would, in the opinion of the investigator and/or medical monitor, place the subject at an unacceptable risk to participate in this study.
* History of or suspected history of alcohol misuse or recreational substance abuse.
* Treatment with oral or IV corticosteroids within 8 weeks prior to screening.
* Concurrent enrolment in another clinical study.
* Receipt of any investigational drug therapy of use of any biologicals within 6 months prior to screening.
* Known history of allergy or reaction to any component of the investigational product.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Piper, MBBS, Study Director — MedImmune Ltd
Locations (4):
- South Africa (3):
  - Research Site, Bloemfontein
  - Research Site, George
  - Research Site, Port Elizabeth
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 participants provided written informed consent and participated in the study at 3 sites in South Africa (2 sites) and the United Kingdom (1 site) between 24Feb2011 and 25Nov2011.
Pre-assignment Details: Eligibile participants in the 10 and 30 mg dose groups received MEDI2338 in an open-label manner. Eligible participants in the 100, 300, and 1000 dose groups were randomized in a 3:1 ratio to receive MEDI2338 or placebo.
Period: Overall Study
Arm/Group | Placebo | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG
Started | 6 (RANDOMIZED SUBJECTS THROUGH STUDY DAY 240-300) | 3 | 3 | 6 | 7 | 6
Completed | 6 | 3 | 3 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Total
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 7 | 6 | 31
Age Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (8.0) | 57.0 (4.0) | 59.7 (11.0) | 60.3 (7.1) | 55.1 (5.3) | 60.8 (6.0) | 59.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 2 | 2 | 0 | 11
  Male | 2 | 2 | 1 | 4 | 5 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 3 | 3 | 6 | 7 | 5 | 6

2. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Clinically Significant Hematology Laboratory Results
Description: Number of participants experiencing clinically significant hematology laboratory results. A clinically significant hematology laboratory result is defined as an abnormal hematology laboratory result that results in a treatment-emergent adverse event.
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Clinically Significant Electrocardiogram Results
Description: Number of participants experiencing clinically significant electrocardiogram results. A clinically significant electrocardiogram result is defined as an abnormal electrocardiogram result that results in a treatment-emergent adverse event.
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Incidence of Clinically Significant Vital Signs Results
Description: Number of participants experiencing clinically significant vital signs results. A clinically significant vital signs result is defined as an abnormal vital signs result that results in a treatment-emergent adverse event.
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Incidence of Clinically Significant Serum Chemistry Laboratory Results
Description: Number of participants experiencing clinically significant serum chemistry laboratory results. A clinically significant serum chemistry laboratory result is defined as an abnormal serum chemistry laboratory result that results in a treatment-emergent adverse event.
Time Frame: Days 1 - 92
Population: All 31 participants entered into the study received MEDI2338 or placebo and were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity
Description: Area under the serum concentration-time curve from time zerio to infinity of MEDI2338
Time Frame: Pre-dose (Day 1) and post-dose (Days 1 [end of infusion, and 30 minutes and 1, 3, 8, and 24 hours postinfusion], 2, 3, 5, 8, 10, 15, 22, 29, 36, 43, 57, 71, and 92)
Population: Of the 31 participants who entered into the study and received MEDI2338 or placebo, 25 participants received only MEDI2338 and were included in the pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: ng x day/mL
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
ng x day/mL | 27550.5 (8163.6) | 104751.1 (40826.2) | 281781.5 (61554.1) | 915668.6 (342545.7) | 3081728.5 (846989.4) |

8. Secondary Outcome: Area Under the Serum Concentration-Time Profile From Time Zero to the Last Measurable Time Point
Description: Area under the serum concentration-time profile from time zero to the last measurable time point of MEDI2338
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng x day/mL
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
ng x day/mL | 24427.8 (8086.4) | 87549.7 (31391.2) | 250155.6 (40613.8) | 846433.3 (303849.8) | 2909818.8 (812729.7) |

9. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI2338
Description: Number of participants with ADA to MEDI2338
Time Frame: Days 1, 57, and 92
Population: Of the 31 participants who entered into the study and received MEDI2338 or placebo, 25 participants received only MEDI2338 and were included in the analysis of ADA
Measure: Number; unit: Participants
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0 |

10. Secondary Outcome: Observed Maximum Concentration (Cmax)
Description: Cmax of MEDI2338
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
ng/mL | 2458.0 (589.1) | 9722.2 (4376.8) | 27122.6 (2845.9) | 106042.5 (23883.9) | 337004.5 (51793.8) |

11. Secondary Outcome: Apparent Terminal Elimination Phase Half-life (t1/2)
Description: t1/2 of MEDI2338
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
Days | 34.85 (5.30) | 40.85 (3.51) | 28.46 (3.37) | 26.76 (5.54) | 24.87 (3.27) |

12. Secondary Outcome: Clearance (CL)
Description: CL of MEDI2338
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/Days
Arm/Group | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 6 | 0
L/Days | 0.387 (0.125) | 0.312 (0.099) | 0.365 (0.071) | 0.360 (0.110) | 0.346 (0.097) |

ADVERSE EVENTS:
Time Frame: Days 1-92
Arm/Group | Placebo | MEDI2338 10 MG | MEDI2338 30 MG | MEDI2338 100 MG | MEDI2338 300 MG | MEDI2338 1000 MG
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 6/6 | 7/7 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | MEDI2338 10 MG (N=3) | MEDI2338 30 MG (N=3) | MEDI2338 100 MG (N=6) | MEDI2338 300 MG (N=7) | MEDI2338 1000 MG (N=6)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.